CLINICAL TRIAL: NCT02267330
Title: A Descriptive Cohort Analysis of Gonadal Radiation Exposure and Risk Secondary to Fluoroscopic Imaging During Trauma Surgery About the Pelvis and Femur
Brief Title: Gonadal Radiation Exposure and Risk Secondary to Fluoroscopic Imaging During Trauma Surgery
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Thomas Higgins, M.D., University of Utah
Other Study IDs: 53129
Record Dates: First submitted 2014-09-03; First posted 2014-10-17 (Estimated); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Hip Fractures; Femur Fractures; Acetabular Fractures; Pelvic Injuries
Keywords: Gonadal Radiation Exposure; Fluoroscopic Imaging; Trauma Surgery; Pelvis fractures; Femur fractures
MeSH Terms: conditions — Hip Fractures; Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Standard of care, Exposure recording: Patient will undergo fracture surgery as per standard of care, and will have radiation exposure recording.
  Interventions: Procedure: Exposure Recording

INTERVENTIONS:
Procedure: Exposure Recording — Patient undergoing fracture surgery will have radiation exposure recorded

SUMMARY:
The aim of this cohort study is to precisely measure patients' exposure to gonadal radiation during orthopaedic trauma surgery involving the acetabulum, pelvis, hip, and femur, and to apply these findings to a previously described and validated formula to determine the increased risk of future adverse health effects to the reproductive organs.

The investigators null hypothesis is standard of care use of x-ray fluoroscopy during treatment of pelvis, hip, and femur fractures will not expose patients to a significant gonadal radiation load. Analysis of patients' intraoperative radiation doses by means of a previously validated formula will not display a significantly increased risk of adverse health events in the reproductive organs.

DETAILED DESCRIPTION:
In the United States, physicians treat more than one and a half million fractures of the pelvis, hip, and femur each year.1-3 Exposure of patients to ionizing radiation during both diagnosis and treatment of these injuries is an unfortunate reality in the standard of care.

Regulations put forth by the US National Radiation Committee (USNRC) include limiting maximum radiation exposure, above background levels, to individual members of the public to less than 1 millisievert (mSv) per year.4 While no current recommendations exist regarding medical exposure in patients, physicians are expected to display judicious practice of both diagnostic and therapeutic procedures during which patients are exposed to ionizing radiation.4 Nevertheless, patients whom undergo trauma activation are exposed to radiation levels that are significant and possibly excessive at 25 to 32 mSv during admission.5,6 The probability that radiation exposure may be reduced is supported by previous studies, which have established that only 60% of surgical trainees take into account the risks of radiation to a patient and that training on intraoperative fluoroscopy technique can decrease patient exposure by more than 50%, while maintaining an equivalent result.7,8

Few previous studies have addressed patient exposure to radiation during operative treatment of orthopaedic injuries.5,9,10 Previous research documenting radiation dose during surgeries of the pelvis and femur have used fluoroscope-calculated dose area product (DAP), which is less accurate than the direct dosimetry proposed in our study.11-13 Furthermore, prior studies have inappropriately determined stochastic risk through the linear no-threshold (LNT) model, which according to the USNRC, provides limited statistical power for epidemiologically based conclusions and overestimates risk at comparatively low doses such as those seen in trauma patients.14,15 Using a more accurate and previously validated model, the stochastic effects of exposure to the reproductive organs can be calculated at a more precise level than provided by previous studies.15,16

The investigators hope this research would allow the orthopaedic community to more accurately express the risks of intraoperative radiation to the patient, while supporting improved training on fluoroscopic technique and promoting the development of less fluoroscopic dependent fixation techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18

Patients with:

* Hip fractures (femoral neck fractures, intertrochanteric fractures)
* Femur fractures (subtrochanteric fractures, femoral shaft fractures)
* Acetabular fractures
* Posterior pelvic ring injuries

Patients requiring surgical fixation of their injuries per standard of care

Exclusion Criteria:

* Any patients under the age of 18
* Any patient not fluent in English.
* Hip fracture undergoing prosthetic replacement

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified for inclusion in the study through routine trauma workup performed at the University of Utah. Patients will be managed through standard of care treatment as dictated by their injuries. If standard of care treatment dictates that a patient requires operative intervention for their injuries and injury pattern is found to meet inclusion criteria, an orthopaedics attending or resident physician will determine the patient's ability to enter the study.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2012-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Gonadal radiation dose | During surgical intervention
  The primary outcome variable will be patient gonadal radiation dose documented through dosimeter application and analysis during standard of care operative intervention.

SECONDARY OUTCOMES:
Fluoroscope-calculated dose. | During surgical intervention
  The investigators will document fluoroscope-calculated dose.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Higgins, M.D., Principal Investigator — University of Utah